CLINICAL TRIAL: NCT06522763
Title: Comparative Randomized, Single Dose, Two-Arm, Parallel Open Label Study to Determine the Bioequivalence of Sulfadoxine/Pyrimethamine 500/25 mg Dispersible Tablet After an Oral Administration to Healthy Adults Under Fasting Conditions
Brief Title: Bioequivalence Study of Sulfadoxine/Pyrimethamine 500/25 mg Dispersible Tablet
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Pharma Nigeria Limited (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUPY-T005
Record Dates: First submitted 2024-07-12; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — Sulfadoxine; Pyrimethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product: 500/25mg Sulfadoxine / Pyrimethamine Dispersible tablets. (Experimental): A single oral dose of 500/25 mg sulfadoxine/pyrimethamine dispersible tablets will be administered.
  Interventions: Drug: Sulfadoxine 500 MG / Pyrimethamine 25 MG dispersible tablets.
- Reference Product: SPAQ-CO® Dispersible tablets. (Active Comparator): A single oral dose of 500/25 mg sulfadoxine/pyrimethamine dispersible tablet from the SPAQ-CO® will be administered.
  Interventions: Drug: Sulfadoxine 500 MG / Pyrimethamine 25 MG dispersible tablets in SPAQ

INTERVENTIONS:
Drug: Sulfadoxine 500 MG / Pyrimethamine 25 MG dispersible tablets. — The 500/25 mg sulfadoxine/pyrimethamine tablet will be dispersed in approximately 10 mL of water in a cup, the mixture obtained will be shaken thoroughly and given immediately to the subject to drink the contents, then the cup will be rinsed with additional approximately 10 mL of water and have the subject drink the contents to assure that the whole dose is taken.
  Arms: Test Product: 500/25mg Sulfadoxine / Pyrimethamine Dispersible tablets.
Drug: Sulfadoxine 500 MG / Pyrimethamine 25 MG dispersible tablets in SPAQ — The 500/25 mg sulfadoxine/pyrimethamine tablet will be dispersed in approximately 10 mL of water in a cup, the mixture obtained will be shaken thoroughly and given immediately to the subject to drink the contents, then the cup will be rinsed with additional approximately 10 mL of water and have the subject drink the contents to assure that the whole dose is taken.
  Arms: Reference Product: SPAQ-CO® Dispersible tablets.

SUMMARY:
The primary objective of this study is to assess the bioequivalence between the test product and the reference product based on Cmax and AUC0->72 for sulfadoxine and pyrimethamine in healthy adults under fasting conditions. The secondary objectives of present study are to describe the Tmax and assess the safety and tolerability profile of both test and reference products.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects male or female (childbearing potential or surgically sterile female (confirmed by medical/operative report or if medical/operative report is not available by ultrasound test)), age 18 to 50 years, inclusive, for post-menopausal female aged between 45 and 65 years inclusive.
2. Body Mass Index (BMI) range8 is within 18.5 - 30.0 Kg/m2.
3. Subject does not have a known allergy to the drug under investigation or any of its ingredients or any other related drugs.
4. Medical history and physical examination within medically acceptable criteria.
5. Subjects having QTc value less than 450 msec for male or less than 440 msec for female at the time of screening.
6. Negative pregnancy test or post-menopausal (ie, at least 1 year without menses and without an alternative medical condition prior to the Screening visit, confirmed by FSH test) if female.
7. Laboratory investigations tests within laboratory reference ranges found in Annex I (ALP and creatinine are accepted if below the reference range after being evaluated by the physician as clinically not significant).
8. Subject is capable of consent.
9. Female subjects of childbearing potential and agrees to use total abstinence or an acceptable contraceptive method of the following: - Systemic contraceptives (birth control pills, injectable/ implantable/ insertable hormonal birth control products, transdermal patch) - Intrauterine device - Condom with intravaginal spermicide

Exclusion Criteria:

1. Medical demographics performed not longer than two weeks before the initiation of the clinical study with significant deviations from the normal ranges
2. Presence of any clinically significant results from laboratory tests found in Annex I, however, ALP and creatinine will be accepted if below reference range after being evaluated by the physician as clinically not significant. Laboratory tests are performed not longer than two weeks before the initiation of the clinical study.
3. History of drug or alcohol abuse.
4. Subject is a heavy smoker (more than 10 cigarettes per day).
5. Subject does not agree to not taking any prescription or non-prescription drugs within at least two weeks before study drug administration and until donating the last sample of the study.
6. Subject does not agree to not taking any vitamins taken for nutritional purposes within at least two days before study drug administration and until donating the last sample of the study.
7. Subject is on a special diet (for example subject is vegetarian).
8. Subject consumes large quantities of alcohol or beverages containing methylxanthines e.g. caffeine (coffee, tea, cola, energy drinks, chocolate etc.).
9. Subject does not agree to not consuming any beverages or food containing alcohol at least 48 hours prior to study drug administration until donating the last sample of the study.
10. Subject does not agree to not consuming any beverages or food containing methylxanthines e.g. caffeine (coffee, tea, cola, energy drinks, chocolate etc.) at least 24 hours prior to the study drug administration until the end of confinement.
11. Subject does not agree to not consuming any beverages or food containing grapefruit at least 7 days prior to study drug administration until donating the last sample of the study.
12. Subject has a history of severe diseases, which have direct impact on the study.
13. Participation in a bioequivalence study or in a clinical study within the last 90 days before study drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Maximal Plasma Concentration (Cmax). | 72 hours
  The confidence intervals of logarithmically transformed Test/Reference ratios for Cmax are set to be within 80.00-125.00% for sulfadoxine and pyrimethamine. ANOVA using 5 % significance level on logarithmically transformed data (with the 90% confidence intervals) of Cmax and AUC0-72 for sulfadoxine and pyrimethamine using WinNonLin statistical software version 8.4 or higher.
Area Under the plasma concentration-time Curve (AUC). | 72 hours
  The confidence intervals of logarithmically transformed Test/Reference ratios for AUC are set to be within 80.00-125.00% for sulfadoxine and pyrimethamine. ANOVA using 5 % significance level on logarithmically transformed data (with the 90% confidence intervals) of AUC0-72 for sulfadoxine and pyrimethamine using WinNonLin statistical software version 8.4 or higher.

SECONDARY OUTCOMES:
Time point of maximal plasma concentration (Tmax) | To be determined within the 72 hours range
  Time of the maximum measured plasma concentration. If the maximum value occurs at more than one time point, Tmax is defined as the first time point with this value.

CONTACTS AND LOCATIONS:
Overall Officials: Majdi Abu Awida, Doctor, Principal Investigator — International Pharmaceutical Research Center ( IPRC)
Locations (1):
- International Pharmaceutical Research Center (IPRC) Queen Rania Street - Sport City Circle,, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The access is controlled, with access only after written approval from IPRC.